CLINICAL TRIAL: NCT06705153
Title: The Effect of Laughter Yoga in Patients with Irritable Bowel Syndrome: a Randomized Controlled Trial
Brief Title: The Effect of Laughter Yoga on Symptom Severity, Depression-anxiety-stress, Sleep Quality and Quality of Life in Patients with Irritable Bowel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ebru BALA, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AtaturkU-EBALA-01
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Laughter Yoga; stress; depression; Anxiety; quality of life; symptom severity; sleep quality
MeSH Terms: conditions — Irritable Bowel Syndrome; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: This randomized controlled study will be conducted to evaluate the effect of laughter yoga in patients with IBS who come to Erzurum City Hospital gastroenterology outpatient clinic. Patient information form, IBS symptom severity score (IBS-SSS), Depression, Anxiety and Stress Scale (DASS-42), Pittsburg Sleep Quality Index (PSQI) and IBS quality of life scale (IBS-QOL) will be applied to the patients. The patients in the intervention group will have laughter yoga for 2 sessions per week (total 8 sessions) for 4 weeks and the patients in the control group will not have laughter yoga. Patients in both groups will be evaluated for IBS-SSS at baseline and at the end of weeks 1, 2, 3 and 4. Patients in both groups will be administered DASS-42, PSQI and IBS-QOL at baseline and at the end of the 4th week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- laughter yoga group (Experimental): The patients in the intervention group will have laughter yoga for 2 sessions per week (total 8 sessions) for 4 weeks in the form of meetings via zoom with the help of a smart cell phone/computer and the patients in the control group will not have laughter yoga. Patients in both groups will be evaluated for IBS-SSS at baseline and at the end of weeks 1, 2, 3 and 4. Patients in both groups will be administered DASS-42, PSQI and IBS-QOL at baseline and at the end of the 4th week. Laughter yoga is a four-part program that lasts about 40 minutes and is led by a leader. These are deep breathing exercises (5-10 minutes), clapping and warm-up exercises (10 minutes), childlike games (10 minutes) and laughter exercises (15 minutes). The philosophy of laughter yoga, a non-invasive and non-pharmacological therapy method that includes breathing techniques that combine unconditional laughter with relaxation and breathing exercises, is based on the statement "movement creates emotion".
  Interventions: Other: laughter yoga
- control group (No Intervention): Patients in the control group will not receive laughter yoga and will use their routine treatment. Patients in both groups will be evaluated for IBS-SSS at baseline and at the end of weeks 1, 2, 3 and 4. Patients in both groups will be administered DASS-42, PSQI and IBS-QOL at baseline and at the end of the 4th week.

INTERVENTIONS:
Other: laughter yoga — Patients who come to the outpatient clinic will be met, informed about the study and written informed consent will be obtained from patients who agree to participate in the study. Patient information form will be applied, baseline measurements will be made (IBS-SSS, DAS-42, PSQI and IBS-QOL) and IBS type will be determined according to Bristol stool scale. Type 1-2 constipation, Type 6-7 diarrhea, Type 1 or Type 2 at the same time with Type 6 or Type 7 will be considered as mixed type IBS and those who do not fit any of the scales will be considered as unclassifiable IBS. A total of 8 sessions will be held with the patients in the intervention group in the form of meetings via zoom with the help of a smart cell phone/computer (2 weekly sessions). The meetings will be in 3 groups.
  Arms: laughter yoga group

SUMMARY:
The study will be conducted to evaluate the effect of laughter yoga on symptom severity, depression, anxiety, stress, sleep and quality of life in patients with Irritable Bowel Syndrome (IBS).

The following hypotheses will be tested in this study:

H1: Laughter yoga reduces symptom severity in patients with IBS. H2: Laughter yoga reduces depression, anxiety and stress in patients with IBS. H3: Laughter yoga improves sleep quality in patients with IBS. H4: Laughter yoga improves quality of life in patients with IBS.

DETAILED DESCRIPTION:
1. Materials and Methods

1.1. Study design and participants This randomized controlled study will be conducted to evaluate the effect of laughter yoga in patients with IBS who come to Erzurum City Hospital gastroenterology outpatient clinic. Patient information form, IBS symptom severity score (IBS-SSS), Depression, Anxiety and Stress Scale (DASS-42), Pittsburg Sleep Quality Index (PSQI) and IBS quality of life scale (IBS-QOL) will be applied to the patients. The patients in the intervention group will have laughter yoga for 2 sessions per week (total 8 sessions) for 4 weeks and the patients in the control group will not have laughter yoga. Patients in both groups will be evaluated for IBS-SSS at baseline and at the end of weeks 1, 2, 3 and 4. Patients in both groups will be administered DASS-42, PSQI and IBS-QOL at baseline and at the end of the 4th week. This work will be conducted in accordance with CONSORT guidelines.

1.2. Sample size and randomization A priori power analysis was calculated in the G. Power 3.1. program to determine the estimated sample size. IBS symptom severity score, the primary measurement tool, was used in power analysis. The sample size was calculated as 50 between two different groups (control group and intervention group) and five measurements (baseline, weeks 1, 2, 3, and 4) with an effect size of Cohen's f = 0.25 (medium effect), power of the test (1-β)=0.95 and α=0.05. Considering the possible losses, 10% drop out was added to the calculated sample and the sample size was calculated as 28 in the intervention group and 28 in the control group, totaling 56.

Patients coming to the outpatient clinic between November-2024 and January-2025 will be determined whether they meet the inclusion criteria. A total of 56 patients will form a sample pool. Potential patients will be numbered in order of arrival at the outpatient clinic. Following the creation of the sample pool, the Random Allocation Software 1.0 program will be used to ensure homogeneous distribution of participants to the groups. In this program, a randomization list will be created with a simple randomization method. In this randomization list, there is a numbered random distribution of 56 participants, 28 in the intervention group and 28 in the control group. Potential participants in the sample pool will be allocated to groups according to the numbers given. 56 patients will be distributed as 28 in the intervention group and 28 in the control group.

1.3. Intervention Patients who come to the outpatient clinic will be met, informed about the study and written informed consent will be obtained from patients who agree to participate in the study. Patient information form will be applied, baseline measurements will be made (IBS-SSS, DAS-42, PSQI and IBS-QOL) and IBS type will be determined according to Bristol stool scale. Type 1-2 constipation, Type 6-7 diarrhea, Type 1 or Type 2 at the same time with Type 6 or Type 7 will be considered as mixed type IBS and those who do not fit any of the scales will be considered as unclassifiable IBS. A total of 8 sessions will be held with the patients in the intervention group in the form of meetings via zoom with the help of a smart cell phone/computer (2 weekly sessions). The meetings will be in 3 groups.

Laughter yoga is a four-part program that lasts about 40 minutes and is led by a leader. These are deep breathing exercises (5-10 minutes), clapping and warm-up exercises (10 minutes), childlike games (10 minutes) and laughter exercises (15 minutes). The philosophy of laughter yoga, a non-invasive and non-pharmacological therapy method that includes breathing techniques that combine unconditional laughter with relaxation and breathing exercises, is based on the statement "movement creates emotion".

Patients in the control group will not receive laughter yoga and will use their routine treatment. At the end of the 1st, 2nd, 3rd and 4th week, IBS-SSS of the patients in the intervention and control groups will be evaluated and at the end of the 4th week, DASS-42, PSQI and IBS-QOL scale will be applied to the patients in both groups.

1.4. Measurement Tools Patient information form, IBS-SSS as the primary measurement tool, DASS-42, PSQI and IBS-QOL scale as secondary measurement tools will be used to collect the data of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with IBS according to Rome IV criteria,
* Scoring 75 and above on the IBS-SSS score,
* DASS-42 scores of 10 and above for depression, 8 and above for anxiety, 15 and above for stress,
* Over 18 years of age,
* Bleeding hemorrhoids, all types of hernia, persistent cough, severe back pain, heart diseases, high blood pressure, urinary incontinence, major psychiatric diseases, pregnancy, cold/flu, no epilepsy, no surgery in the last three months, etc.
* Patients with a smartphone/computer where it is possible to participate in a video call for laughter yoga,
* Patients without communication problems and
* Patients who agree to participate in the study will be included in the study.

Exclusion Criteria:

* who do not practice laughter yoga,
* who do not attend regularly,
* Patients whose treatment regimen has changed and
* Patients who wish to leave the study will be excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female and male
Enrollment: 56 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-01-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
IBS Symptom Severity Score - (IBS-SSS) | IBS-SSS will be assessed 5 times in total, at baseline and weeks 1, 2, 3 and 4.
  The IBS-SSS will be used as the primary measurement tool. The scale is used to assess the course of the disease and the treatment process. The IBS-SSS assesses the severity and duration of abdominal pain, complaints of abdominal bloating, distension, fullness and gas, satisfaction with bowel habits and how bowel symptoms affect a person's life. Each of the scale items consists of a total of 5 questions ranging from 0 to 100 points. The scale score ranges from 0 to 500, with higher scores indicating increased symptom severity. In the scale, 0-74 points are classified as remission, 75-174 as mild, 175-299 as moderate, and 300 points and above as severe severe IBS. The assessment states that a 50-point reduction is sufficient for clinical improvement. The IBS-SSS was chosen as the primary measurement tool because it is effective in evaluating the course of IBS and the effectiveness of treatment and is widely used.

SECONDARY OUTCOMES:
Depression-Anxiety-Stress Scale (DASS-42) | DASS-42 will be evaluated 2 times in total, at baseline and week 4.
  Secondary measuring instrument: DASS-42 will be used. The scale is 4-point Likert-type and consists of 3 sub-dimensions (depression, anxiety, stress). Each sub-dimension has 14 items and the scale has 42 items in total. Each of the depression, anxiety and stress scores ranged from 0 to 42, with depression, anxiety and stress increasing as the score increased. Depression was divided into 5 categories as remission (0-9), mild (10-13), moderate (14-20), advanced (21-27) and very advanced (28-42); anxiety remission (0-7), mild (8-9), moderate (10-14), advanced (15-19) and very advanced (20-42); and stress remission (0-14), mild (15-18), moderate (19-25), advanced (26-33) and very advanced (34-42).
Pittsburg Sleep Quality Index (PSQI) | PSQI will be evaluated 2 times in total, at baseline and week 4.
  Secondary measurement tool: PSQI will be used. The scale consists of 24 questions. 19 of the questions were self-assessment questions. Five questions are answered by the individual's spouse or a friend. These five questions are used for clinical information and are not included in the scoring. Self-assessment questions include various factors related to sleep quality. The 18 scored items were grouped into 7 component scores. Some of the components consist of a single substance, while others are obtained by grouping several substances. Each item is evaluated with a score between 0-3.The scores of the 7 components of the scale are calculated and summed to obtain a total scale score. A high total scale score indicates poor sleep quality. The scale indicates the presence or absence of sleep disorders or the prevalence of sleep disorders. A PSQI total scale score of 5 and above indicates poor sleep quality.
Irritable Bowel Syndrome Quality of Life Scale (IBSQOL) | The IBS-QOL scale will be evaluated 2 times in total, at baseline and week 4.
  The IBS-QOL scale will be used as the other secondary measurement tool. The scale prepared for IBS patients is 5-point Likert-type and consists of a total of 34 items and 8 sub-dimensions. Scale sub-dimensions are dysphoria, activity, body image, health anxiety, food avoidance, social reaction, sexual and social relationship. The total score of the scale is obtained by summing the scores obtained from 34 items, and the sub-dimension scores are obtained by summing each of the sub-dimensions separately. The sub-dimension and total scores of the IBS-QOL scale range between 0-100. Higher scale scores indicate a decreased quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum City Hospital, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes